CLINICAL TRIAL: NCT01769534
Title: Prospective Registry and Cystic Fluid Banking for Patients Undergoing EUS-FNA for the Evaluation of Pancreatic Cystic Lesions.
Brief Title: Registry and Fluid Banking of Pancreatic Cystic Lesions
Status: Terminated | Type: Observational
Why Stopped: Administratively inactivated
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: 2487
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Pancreatic Cysts
MeSH Terms: conditions — Pancreatic Cyst

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Pancreatic cyst fluid
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to follow patients, who have small mucinous cysts in the pancreas, prospectively over a 5-year period.

DETAILED DESCRIPTION:
The patients will present to our endoscopy unit for EUS-FNA to work up pancreatic cystic lesion(s). At that time, we will recruit them to be in the patient registry and tissue repository. Their enrollment in the patient registry will allow us to contact them annually for survey purposes. Their enrollment in the tissue repository will allow us to store left-over pancreatic cyst fluid that was already aspirated for analysis (as part of the standard-of-care workup for pancreatic cysts).

ELIGIBILITY:
Inclusion Criteria:

* consented patients between age 18 to 85 who are referred for EUS evaluation of pancreatic cysts.

Exclusion Criteria:

* Patient unable to give informed consent
* age<18 or >85, patients with clinically suspected pseudocysts.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients will present to our endoscopy unit for EUS-FNA to work up pancreatic cystic lesion(s).
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2012-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
To validate the Sendai criteria prospectively in patients with pancreatic cysts. | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: John T Maple, M.D., Principal Investigator — University of Oklahoma
Locations (1):
- Endoscopy Centrer at OU Medical Center, Oklahoma City, Oklahoma, United States